CLINICAL TRIAL: NCT03975920
Title: The Restful Jaw Device: A New Way to Support and Protect the Jaw During Third Molar Extractions
Brief Title: Assessing a New Jaw Support Device During Third Molar Extractions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: HealthPartners Institute (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DENT-2019-27811; 4R44DE026663-02 (NIH)
Record Dates: First submitted 2019-05-21; First posted 2019-06-05 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Impacted Third Molar Tooth; Temporomandibular Disorder
Keywords: jaw support device; wisdom teeth; impacted; Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders; Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: In this two-arm parallel randomized clinical trial (RCT) design, 294 patients undergoing 3rd molar extractions with moderate/deep sedation or general anesthesia will be randomly allocated to Usual Care (UC) or Experimental Care (EC). The study intervention for EC is use of the Restful Jaw version 2 (RJ2) device, which supports the jaw during the extractions, with concurrent use of a bite block. The study control is UC, which involves the dental assistant supporting the jaw during the extractions with concurrent use of a bite block.
Who Masked: Investigator
Masking Description: In this RCT, it is not feasible to blind patients, surgeons, or dental assistants to treatment after the intervention assignments have occurred, so they will not be blinded. It is, however, feasible to mask the sequence of treatment assignments until the moment each assignment is made, and this will be done, as described in Section 5.4.1, above.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Usual Care (UC) (No Intervention): The study control is UC, which involves the dental assistant supporting the jaw during the extractions with concurrent use of a bite block.
- Experimental Care (EC) (Experimental): The study intervention for EC is use of the Restful Jaw version 2 (RJ2) device, which supports the jaw during the extractions, with concurrent use of a bite block.
  Interventions: Device: The Restful Jaw Device

INTERVENTIONS:
Device: The Restful Jaw Device — The Restful Jaw Device is used to support the jaw during dental procedures including surgical removal of 3rd molars (wisdom teeth) with sedation. The device is designed to counter the downward forces placed on the mandible by clinicians during dental procedures and prevent jaw hyperextension (opening too wide) while providing a secure, stable jaw position. When 3rd molar teeth are surgically removed with sedation, a dental assistant stands behind the dental chair and supports the patient's jaw with both hands under the patient's jaw. This device replicates the dental assistant in holding the jaw during dental procedures.
  Other Names: RJ2
  Arms: Experimental Care (EC)

SUMMARY:
During mandibular 3rd molar (wisdom tooth) extractions, when a downward force is placed on the patient's jaw, the patient must tense his/her jaw muscles to oppose it. Patients under moderate/deep sedation or general anesthesia cannot tense their muscles to counter this downward force to prevent injury to the jaw including the temporomandibular joint (TMJ). Bite blocks hold the patient's mouth open but do not counter this downward force on the mandible. Currently, oral and maxillofacial surgeons (OMSs) when surgically removing 3rd molars (wisdom teeth) with moderate/deep sedation or general anesthesia have a dental assistant that stands behind the chair and places their hands on both sides of the jaw to support it and oppose the downward force on the patient's jaw during the extractions. It is hard for the dental assistant to maintain support while anticipating the direction and amount of force placed by the OMS on the patient's jaw during the surgical removal. This may explain the finding that almost a quarter of new onset TMD cases in young adults is associated with 3rd molar removal. This study will look at the use of a jaw support device to provide a stable counterforce to downward forces on the jaw, thus preventing jaw hyperextension and injury to the jaw.

DETAILED DESCRIPTION:
Dental procedures can cause jaw pain, discomfort and fatigue from opening the mouth too long or too wide, or by placing too much force on the jaw. (1-15) Opening too wide can also cause hyperextension of the jaw. During and after long dental procedures, patients frequently report jaw pain, fatigue, or discomfort. This pain and dysfunction characterizes temporomandibular disorders (TMD), which can be short-term or may become chronic. TMD occurrence is frequently associated with trauma from dental procedures, including 3rd molar extractions. (1-15) Also, dental procedures may aggravate pre-existing subclinical TMD symptoms. (16)

When a downward force is placed on the patient's jaw to surgically remove the mandibular (lower) 3rd molars, the patient must tense his/her jaw muscles to oppose it. This can result in jaw pain, discomfort or fatigue, especially if the force is high or prolonged. Patients under moderate/deep sedation or general anesthesia cannot tense their muscles to counter this downward force to prevent injury to the jaw. Bite blocks hold the patient's mouth open but do nothing to counter this downward force on the jaw. Opening a patient's mouth too wide can cause jaw hyperextension; a long extraction procedure time can also lead to injury of the jaw. Currently, oral and maxillofacial surgeons (OMSs) when surgically removing 3rd molars (wisdom teeth) with moderate/deep sedation or general anesthesia have at least 2 dental assistants present. The first dental assistant provides suction and gives the surgical instruments to the surgeon. The second dental assistant is a certified anesthesia dental assistant who monitors the patient's vitals as well as oxygen and carbon dioxide levels while providing the patient with medications intravenously. This second dental assistant also inserts the bite block and then stands behind the chair and places their hands on both sides of the jaw to support it and oppose the downward force on the patient's jaw during the extractions. If additional intravenous medications are needed during the surgery, the surgery has to stop (lost time) and the OMS or the first dental assistant supports the jaw until the second dental assistant completes the medication administration. Based on clinical experience, the second dental assistant often experiences fatigue and pain in their hands, arms, neck and shoulders during long or difficult procedures, which can affect his/her ability to support the jaw. Given the second dental assistant's many duties and responsibilities, it is hard for the assistant to provide constant good jaw support while anticipating the direction and amount of force placed by the OMS on the patient's jaw during 3rd molar surgical removal. This may explain the finding that almost a quarter of new onset of TMD cases in young adults is associated with 3rd molar removal. This patient safety issue can be addressed during 3rd molar surgical removal by using a bite block to hold the mouth open and concurrently using a jaw support device under the jaw to provide a stable counter force to downward forces on the jaw, thus preventing jaw hyperextension and injury to the jaw. This would also free the second dental assistant from holding the jaw so he/she can concentrate on his/her other duties, which would improve patient safety.

In this two-arm parallel randomized clinical trial design, 294 patients undergoing 3rd molar extractions with moderate/deep sedation or general anesthesia will be randomly allocated to Usual Care (UC) or Experimental Care (EC).

Patients presenting for surgical removal of 3rd molars will be invited to participate in the study at the time of their oral surgery consult. The OMS will determine if the patient meets eligibility criteria, explain the study and invite them to participate. At the time of 3rd molar removal, the OMS and their dental assistants will follow their standard procedures for obtaining consent from patients for 3rd molar removal with moderate/deep sedation. In addition, they will confirm the patient's interest to participate in the study, ask if they have any questions an obtain consent. The jaw device will be placed for those who are randomized into the EC group. The OMS will follow their standard protocol for removal of the teeth. The only change will be that the dental assistant standing behind the chair will be present at all time to readjust the device position as needed or remove the device as indicated. The default in the case of device malfunction is for the device to fall away from the patient and the dental assistant will be immediately available to take over supporting the patient's jaw with their hands, which is one of their standard responsibilities when the device is not used.

Patients will report temporomandibular disorders (TMD) pain via questionnaires at baseline and at the 1-, 3-, and 6-month follow-up time points via email, phone and/or text.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 to 30 years of age at time of enrollment;
* Willing to provide informed consent to be randomized to either using the device or not when having surgical removal of 3rd molars with moderate/deep sedation or general anesthesia;
* Requires surgical removal of bilateral mandibular 3rd molars with moderate/deep sedation or general anesthesia; concurrent maxillary 3rd molars removal allowed;
* American Society of Anesthesiologists (ASA) Physical Status category 1 (normal healthy patient) or Category 2 (patient with mild systemic disease);
* Available to be contacted for study purposes by e-mail, phone and/or text;
* Willing to provide contact information for one other person who will know the patient's whereabouts in the event the patient cannot be reached. This contact information must be different from the patient's contact information;
* Willing to comply with all study procedures and be available for the six month duration of data collection.

Exclusion Criteria:

* In the past 3 months, reports the presence of TMD pain in their temples, jaw joints or jaw muscles;
* Contraindication(s) for moderate/deep sedation or general anesthesia;
* Any condition or situation the surgeon determines that would prevent the patient from participating in this study;
* Inability to understand study procedures or provide consent in English;
* Device does not fit mandible;
* Supernumerary 3rd molars present.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Schiffman, DDS, MS, Principal Investigator — University of Minnesota
Locations (4):
- United States (4):
  - Metro Dentalcare Specialty Center, Burnsville, Minnesota
  - HealthPartners Eden Prairie Clinc, Eden Prairie, Minnesota
  - University of Minnesota School of Dentistry, Minneapolis, Minnesota
  - HealthPartners Como Clinic, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
To facilitate the conduct of further analyses with the data we collect, we will create Limited Data Sets from the completed project in a manner consistent with human subject protection and HIPAA privacy regulations.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication of the first paper.
Access Criteria: These resources will be available to the NIDCR or to other approved investigators according to requirements imposed by the governing IRB and legal requirements, including HIPAA and Data Use Agreements.

REFERENCES:
- [Background] Friedman JW. The prophylactic extraction of third molars: a public health hazard. Am J Public Health. 2007 Sep;97(9):1554-9. doi: 10.2105/AJPH.2006.100271. Epub 2007 Jul 31. PMID 17666691
- [Background] Huang GJ, Rue TC. Third-molar extraction as a risk factor for temporomandibular disorder. J Am Dent Assoc. 2006 Nov;137(11):1547-54. doi: 10.14219/jada.archive.2006.0090. PMID 17082281
- [Background] Huang GJ, Cunha-Cruz J, Rothen M, Spiekerman C, Drangsholt M, Anderson L, Roset GA. A prospective study of clinical outcomes related to third molar removal or retention. Am J Public Health. 2014 Apr;104(4):728-34. doi: 10.2105/AJPH.2013.301649. Epub 2014 Feb 13. PMID 24524521
- [Background] Huang GJ, Drangsholt MT, Rue TC, Cruikshank DC, Hobson KA. Age and third molar extraction as risk factors for temporomandibular disorder. J Dent Res. 2008 Mar;87(3):283-7. doi: 10.1177/154405910808700313. PMID 18296615
- [Background] Huang GJ, LeResche L, Critchlow CW, Martin MD, Drangsholt MT. Risk factors for diagnostic subgroups of painful temporomandibular disorders (TMD). J Dent Res. 2002 Apr;81(4):284-8. doi: 10.1177/154405910208100412. PMID 12097315
- [Background] Juhl GI, Jensen TS, Norholt SE, Svensson P. Incidence of symptoms and signs of TMD following third molar surgery: a controlled, prospective study. J Oral Rehabil. 2009 Mar;36(3):199-209. doi: 10.1111/j.1365-2842.2008.01925.x. PMID 19207447
- [Background] Akhter R, Hassan NM, Ohkubo R, Tsukazaki T, Aida J, Morita M. The relationship between jaw injury, third molar removal, and orthodontic treatment and TMD symptoms in university students in Japan. J Orofac Pain. 2008 Winter;22(1):50-6. PMID 18351034
- [Background] Velly AM, Gornitsky M, Philippe P. Contributing factors to chronic myofascial pain: a case-control study. Pain. 2003 Aug;104(3):491-499. doi: 10.1016/S0304-3959(03)00074-5. PMID 12927621
- [Background] Okeson JP. Bell's orofacial pains: The clinical management of orofacial pain, sixth edition. Vol 6. Illinois: Quintessence Publishing; 2005.
- [Background] Pullinger AG, Monteiro AA. History factors associated with symptoms of temporomandibular disorders. J Oral Rehabil. 1988 Mar;15(2):117-24. doi: 10.1111/j.1365-2842.1988.tb00760.x. PMID 3163728
- [Background] LeResche L, Mancl LA, Drangsholt MT, Huang G, Von Korff M. Predictors of onset of facial pain and temporomandibular disorders in early adolescence. Pain. 2007 Jun;129(3):269-278. doi: 10.1016/j.pain.2006.10.012. Epub 2006 Nov 28. PMID 17134830
- [Background] Plesh O, Gansky SA, Curtis DA, Pogrel MA. The relationship between chronic facial pain and a history of trauma and surgery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1999 Jul;88(1):16-21. doi: 10.1016/s1079-2104(99)70187-3. PMID 10442939
- [Background] Butler JH, Folke LE, Bandt CL. A descriptive survey of signs and symptoms associated with the myofascial pain-dysfunction syndrome. J Am Dent Assoc. 1975 Mar;90(3):635-9. doi: 10.14219/jada.archive.1975.0147. PMID 1054051
- [Background] Fricton JR, Kroening R, Haley D, Siegert R. Myofascial pain syndrome of the head and neck: a review of clinical characteristics of 164 patients. Oral Surg Oral Med Oral Pathol. 1985 Dec;60(6):615-23. doi: 10.1016/0030-4220(85)90364-0. PMID 3865133
- [Background] Sahebi S, Moazami F, Afsa M, Nabavi Zade MR. Effect of lengthy root canal therapy sessions on temporomandibular joint and masticatory muscles. J Dent Res Dent Clin Dent Prospects. 2010 Summer;4(3):95-7. doi: 10.5681/joddd.2010.024. Epub 2010 Sep 16. PMID 22991607
- [Background] Humphrey SP, Lindroth JE, Carlson CR. Routine dental care in patients with temporomandibular disorders. J Orofac Pain. 2002 Spring;16(2):129-34. PMID 12043519
- [Background] American Association of Oral and Maxillofacial Surgeons. Parameters of care: Clinical and practice guidelines for oral and maxillofacial surgeons. 2012. Available at http://www.mfch.cz/doc/ParCare2012Complete.pdf
- [Background] Fernandes P, Velly AM, Anderson GC. A randomized controlled clinical trial evaluating the effectiveness of an external mandibular support device during dental care for patients with temporomandibular disorders. Gen Dent. 2013 Sep-Oct;61(6):26-31. PMID 24064159
- [Background] Zucuskie T. A controlled clinical trial of the usefulness of an external mandibular support device during routine dental care. Minneapolis: University of Minnesota; 1996.
- [Background] Schiffman EL, Look JO, Hodges JS, Swift JQ, Decker KL, Hathaway KM, Templeton RB, Fricton JR. Randomized effectiveness study of four therapeutic strategies for TMJ closed lock. J Dent Res. 2007 Jan;86(1):58-63. doi: 10.1177/154405910708600109. PMID 17189464
- [Background] Lan KKG, DeMets DL. Design and analysis of group sequential tests based on the type 1 error spending rate function. Biometrika. 1987;74:149- 154.
- [Background] Gonzalez YM, Schiffman E, Gordon SM, Seago B, Truelove EL, Slade G, Ohrbach R. Development of a brief and effective temporomandibular disorder pain screening questionnaire: reliability and validity. J Am Dent Assoc. 2011 Oct;142(10):1183-91. doi: 10.14219/jada.archive.2011.0088. PMID 21965492
- [Derived] Uppgaard R, Nadeau R, Schiffman EL, Stiharu T, Johnson KS, Hodges JS, Velly AM. Occurrence and Predictors of Postoperative Preauricular and Masticatory Muscle Pain Symptoms After Surgical Removal of Third Molars: A Single-Blind Randomized Controlled Trial Comparing Dental Assistants Supporting the Mandible and the Restful Jaw Device. J Oral Maxillofac Surg. 2024 Jan;82(1):6-18. doi: 10.1016/j.joms.2023.09.021. Epub 2023 Oct 5. PMID 37898152

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at an academic institution, 2 clinics that are a part of a large group practice, and a clinic in the community between June 2019 and August 2020. The first participant was enrolled on June 25, 2019 and the last participant was enrolled on August 27, 2020.
Pre-assignment Details: A total of 180 participants were enrolled through consult and surgical appointments for removal of wisdom teeth. Nine (9) participants were not randomized due to change in anesthesia or were unable to complete their procedure prior to enrollment closure. 171 participants were randomized into the study; of those, 2 were removed from the study due to protocol deviations (determined did not meet inclusion criteria).
Groups:
- Usual Care (UC): The study control is Usual Care (UC), which involves the dental assistant supporting the jaw during the extractions with concurrent use of a bite block.
- Experimental Care (EC): The study intervention for Experimental Care (EC) is use of the Restful Jaw version 2 (RJ2) device, which supports the jaw during the extractions, with concurrent use of a bite block.
  The Restful Jaw Device: The Restful Jaw Device is used to support the jaw during dental procedures including surgical removal of 3rd molars (wisdom teeth) with sedation. The device is designed to counter the downward forces placed on the mandible by clinicians during dental procedures and prevent jaw hyperextension (opening too wide) while providing a secure, stable jaw position. When 3rd molar teeth are surgically removed with sedation, a dental assistant stands behind the dental chair and supports the patient's jaw with both hands under the patient's jaw. This device replicates the dental assistant in holding the jaw during dental procedures.
Period: Overall Study
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Started | 84 (Due to inclusion criteria protocol deviation, data from 1 participant was not used in the analysis.) | 87 (Due to inclusion criteria protocol deviation, data from 1 participant was not used in the analysis.)
1-Month Follow-up Survey | 80 | 85
3-Month Follow-up Survey | 78 | 84
6-Month Follow-up Survey | 80 | 83
Completed | 80 | 83
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Did not complete survey | 2 | 1

BASELINE CHARACTERISTICS:
Population: One (1) protocol deviation occurred in the Usual Care group and one (1) protocol deviation occurred in the Experimental group that required removal of their data; patients did not meet the inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (UC) | Experimental Care (EC) | Total
Number analyzed (Participants) | 83 | 86 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 83 | 86 | 169
  >=65 years | 0 | 0 | 0
Age, Customized [Count of Participants; unit: Participants]
  18-30 years | 83 | 86 | 169
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 57 | 109
  Male | 31 | 29 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 11 | 15
  Not Hispanic or Latino | 74 | 66 | 140
  Unknown or Not Reported | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 6 | 13 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 57 | 55 | 112
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 83 | 86 | 169

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Pain at Follow-up With Wide Opening, or Pain in the Temple, Jaw Joint or Jaw Muscles.
Description: The primary outcome is the self-report of the occurrence of TMD pain post-baseline. All subjects were pain-free at baseline (i.e., pre-surgically) for TMD pain. TMD pain is deemed to have occurred if the subject's self report endorses at 1, 3 or 6 months post-baseline either or both of the following questions: 1. Pain in jaw when opening mouth wide or 2. Pain in temples, jaw joints or jaw muscles.
Time Frame: 1 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 80 | 85
Participants
  Pain reported at 1 month | 26 | 32
  No pain reported at 1 month | 54 | 53

2. Primary Outcome: Occurrence of Pain at Follow-up With Wide Opening, or Pain in the Temple, Jaw Joint or Jaw Muscles.
Description: as for outcome 1
Time Frame: 3 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 78 | 84
Participants
  Pain reported at 3 months | 18 | 21
  No pain reported at 3months | 60 | 63

3. Primary Outcome: Occurrence of Pain at Follow-up With Wide Opening, or Pain in the Temple, Jaw Joint or Jaw Muscles.
Description: as for outcome 1
Time Frame: 6 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 80 | 83
Participants
  Pain reported at 6 months | 16 | 21
  No pain reported at 6 months | 64 | 62

4. Secondary Outcome: Occurrence of Pain Related TMD at Follow-up Using the TMD Pain Screener Questionnaire.
Description: The occurrence of TMD pain post-baseline will be measured using the reliable and valid TMD Pain Screener Questionnaire. This subject self-report measure is comprised of 3 questions assessing the duration of TMD pain, presence of jaw pain or stiffness upon awakening, and activities that change TMD pain. TMD pain is deemed to have occurred if the subject's self report at 1, 3 or 6 months post-baseline is positive for the presence of TMD pain per the TMD Pain Screener.
Time Frame: 1 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 79 | 83
Participants
  Pain reported at 1 month | 17 | 18
  No pain reported at 1 month | 62 | 65

5. Secondary Outcome: Occurrence of Pain Related TMD at Follow-up Using the TMD Pain Screener Questionnaire.
Description: as for outcome 4
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 78 | 82
Participants
  Pain reported at 3 months | 7 | 8
  No pain reported at 3 months | 71 | 74

6. Secondary Outcome: Occurrence of Pain Related TMD at Follow-up Using the TMD Pain Screener Questionnaire.
Description: as for outcome 4
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 80 | 80
Participants
  Pain reported at 6 months | 6 | 5
  No pain reported at 6 months | 74 | 75

7. Secondary Outcome: Intensity of Pain at Follow-up Using the Characteristic Pain Index (CPI).
Description: Subjects will compete at 1, 3 or 6 months post-baseline the reliable and valid Characteristic Pain Index (CPI) that measures pain intensity. It is comprised of 3 items assessed using numerical rating scales (0-10): current pain, worst pain and average pain. The final score is the average of these 3 items x 10. The CPI is part of the Graded Chronic Pain Scale (GCPS).
Time Frame: 1 Month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 80 | 85
score on a scale | 8.2 (1.8) | 10.2 (1.8)

8. Secondary Outcome: Intensity of Pain at Follow-up Using the Characteristic Pain Index (CPI).
Description: as for outcome 7
Time Frame: 3 Months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 78 | 84
score on a scale | 3.6 (1.4) | 5.5 (1.3)

9. Secondary Outcome: Intensity of Pain at Follow-up Using the Characteristic Pain Index (CPI).
Description: as for outcome 7
Time Frame: 6 Months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 80 | 83
score on a scale | 2.5 (1.1) | 4.9 (1.0)

10. Secondary Outcome: Occurrence of TMJ Noise at Follow-up Using Self Report.
Description: TMJ noise is deemed to have occurred at 1, 3 or 6 months post-baseline if the subject's self report endorses the question: Have you had any clicking or popping in your jaw joints?
Time Frame: 1 Month
Population: The flow chart numbers for the overall study indicate participants' completion as reported for the primary outcome. The numbers represented here indicate that all participants randomized into the study did not complete all of the questions to calculate this secondary outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 79 | 85
Participants
  TMJ noise reported at 1 month | 5 | 12
  No TMJ noise reported at 1 month | 74 | 73

11. Secondary Outcome: Occurrence of TMJ Noise at Follow-up Using Self Report.
Description: as for outcome 10
Time Frame: 3 Months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 77 | 82
Participants
  TMJ noise reported at 3 months | 9 | 12
  No TMJ noise reported at 3 months | 68 | 70

12. Secondary Outcome: Occurrence of TMJ Noise at Follow-up Using Self Report.
Description: as for outcome 10
Time Frame: 6 Months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 79 | 83
Participants
  TMJ noise reported at 6 months | 12 | 15
  No TMJ noise reported at 6 months | 67 | 68

13. Secondary Outcome: Change in Jaw Pain at Follow-up Using Self-report.
Description: Subjects will report any change in jaw pain at 1, 3 or 6 months post-baseline using this question: How would you describe the change (if any) in your jaw pain since it started? The response options are: Much Worse (1), Slightly Worse(2), No Change(3), Slightly Better(4) or Much Better(5).
Time Frame: 1 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 80 | 85
Participants
  Change in jaw pain from baseline much better; self-report | 19 | 16
  Change in jaw pain from baseline slightly better; self-report | 4 | 7
  No change in jaw pain from baseline; self-report | 2 | 7
  Change in jaw pain from baseline slightly worse; self-report | 0 | 1
  Change in jaw pain from baseline much worse; self-report | 1 | 1
  No jaw pain reported | 54 | 53

14. Secondary Outcome: Change in Jaw Pain at Follow-up Using Self-report.
Description: as for outcome 13
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 77 | 84
Participants
  Change in jaw pain from baseline much better; self-report | 8 | 9
  Change in jaw pain from baseline slightly better; self-report | 3 | 4
  No change in jaw pain from baseline; self-report | 5 | 5
  Change in jaw pain from baseline slightly worse; self-report | 1 | 2
  Change in jaw pain from baseline much worse; self-report | 0 | 1
  No pain reported | 60 | 63

15. Secondary Outcome: Change in Jaw Pain at Follow-up Using Self-report.
Description: as for outcome 13
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Experimental Care (EC)
Number analyzed (Participants) | 80 | 83
Participants
  Change in jaw pain from baseline much better; self-report | 7 | 8
  Change in jaw pain from baseline slightly better; self-report | 0 | 4
  No change in jaw pain from baseline; self-report | 8 | 8
  Change in jaw pain from baseline slightly worse; self-report | 1 | 1
  Change in jaw pain from baseline much worse; self-report | 0 | 0
  No pain reported | 64 | 62

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: By definition, no Serious Adverse Events, All-Cause Mortality, and Other (Not Including Serious) Adverse Events occurred in this study.
Arm/Group | Usual Care (UC) | Experimental Care (EC)
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/87
Other Adverse Events (participants affected / at risk) | 0/84 | 0/87

LIMITATIONS AND CAVEATS:
Limitations include that outcomes were self-reported, and patients were not examined at follow-up. Enrollment was impacted by stopping of patient recruitment at the beginning of the COVID pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT03975920/Prot_SAP_002.pdf
  • Informed Consent Form (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT03975920/ICF_001.pdf